CLINICAL TRIAL: NCT02734966
Title: A Multi-center, Randomized, Double-blind, Active Control Phase II Study to Investigate Multiple Dosage and Treatments of Magnesium Isoglycyrrhizinate Injection to Cure the Acute Drug-induced Liver Injury
Brief Title: Efficacy and Safety Study of Magnesium Isoglycyrrhizinate Injection in Subjects With Acute Drug-induced Liver Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZTDQ01341301
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Drug-Induced Liver Injury
Keywords: Drug-Induced; Acute Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — 18alpha,20beta-hydroxy-11-oxo-norolean-12-en-3beta-yl-2-O-beta-D-glucopyranurosyl-alpha-D-glucopyranosiduronate magnesium tetrahydrate; Long-Term Synaptic Depression; Tiopronin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- arm 1 (Experimental): lower dose： Magnesium Isoglycyrrhizinate injection 100mg OD for 4 weeks
  Interventions: Drug: Magnesium Isoglycyrrhizinate Injection 100mg OD
- arm 2 (Experimental): higher dose：Magnesium Isoglycyrrhizinate injection 200mg OD for 4 weeks.
  Interventions: Drug: Magnesium Isoglycyrrhizinate Injection 200mg OD
- Tiopronin Injection (Active Comparator): Tiopronin Injection 200mg OD for 4 weeks
  Interventions: Drug: Tiopronin Injection

INTERVENTIONS:
Drug: Magnesium Isoglycyrrhizinate Injection 100mg OD — Magnesium Isoglycyrrhizinate Injection 100mg OD
  Other Names: Jiangsu Chia Tai Tianqing Pharmaceutical Group Co., Ltd.
  Arms: arm 1
Drug: Magnesium Isoglycyrrhizinate Injection 200mg OD — Magnesium Isoglycyrrhizinate Injection 200mg OD for 4 weeks
  Other Names: Jiangsu Chia Tai Tianqing Pharmaceutical Group Co., Ltd.
  Arms: arm 2
Drug: Tiopronin Injection — Tiopronin Injection 200mg OD
  Other Names: Jinan Limin Pharmaceutical Co., Ltd.
  Arms: Tiopronin Injection

SUMMARY:
The purpose of this study is to investigate the safety, effective dosage and treatment of Magnesium Isolycyrrhizinate Injection to cure the acute drug-induced liver injury compared with the Tiopronin Injection.

DETAILED DESCRIPTION:
The pharmacology research shows that Magnesium Isoglycyrrhizinate could significantly decrease the elevation of ALT and AST coursed by carbon tetrachloride, D-galactosamine and Thioacetamide. It could also significantly reduce the injury on the liver coursed by D-galacosamine and immunologic factors. Magnesium Isoglycyrrhizinate with strong anti-inflammatory effect could protect the liver cell and improve the liver function.

ELIGIBILITY:
Inclusion Criteria:

* RACUM ≥6
* ALTs ≥2ULN, but TBiL is ≤ 3 ULN.It may be associated with AST or ALP or TBiL exceed the upper limit of normal
* Liver biochemical abnormalities duration of no more than three months
* Patients need to fully understand and sign the inform consent form.

Exclusion Criteria:

* The liver injury is caused by other diseases, such as virus hepatitis, alcohol and non-alcohol fatty liver disease or the autoimmune liver disease.
* The patients with the acute hepatic failure or hepatic decompensation, such as hepatic encephalopathy, ascites, albumin is ≤ 35g/L, prothrombin time is elongated more than 2 seconds compared to its normal range.
* The value of the TBiL is > 3ULN.
* The value of serum creatinine is > 1.5ULN.
* Patients who have severe organic diseases on heart, lungs, brain, kidney and gastrointestinal tract.
* Patients who are taking the drugs that might interfere the trial.
* Patients who are allergic or intolerant to the study drug.
* Patients who are not able to express the chief complaint, for example, the patients with psychosis and severe neurosis.
* Patients who are compliant with protocol.
* Women who are pregnant, breast-feeding or with childbearing potential.
* Patients who have attended other clinical trials within 3 months.
* Not appropriate to be included after assessing by the investigators.

ULN=Upper Limited Normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rate of ALT normalization at week 4 of treatment | 4 weeks

SECONDARY OUTCOMES:
rates of ALT normalization at weeks 1, 2, and 3 of treatment | 3 weeks
change of ALT at weeks 1, 2, 3 and 4 of treatment; | 4 weeks
change of AST at weeks 1, 2, 3 and 4 of treatment. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minde Zeng, MD, Principal Investigator — RenJi Hospital
Locations (8):
- China (8):
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Nanjing Pulmonary Hospital, Nanjing, Jiangsu
  - 85 Hospital of People's Liberation Army, Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Integrated Chinese and Western Medicine Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maria VA, Victorino RM. Development and validation of a clinical scale for the diagnosis of drug-induced hepatitis. Hepatology. 1997 Sep;26(3):664-9. doi: 10.1002/hep.510260319. PMID 9303497
- [Background] Watkins PB, Seeff LB. Drug-induced liver injury: summary of a single topic clinical research conference. Hepatology. 2006 Mar;43(3):618-31. doi: 10.1002/hep.21095. PMID 16496329